CLINICAL TRIAL: NCT04371926
Title: Prophylactic Benefit of Hydroxychloroquine in COVID-19 Cases With Mild to Moderate Symptoms and in Healthcare Workers With High Exposure Risk (PREVENT)
Brief Title: Prophylactic Benefit of Hydroxychloroquine in COVID-19 Cases With Mild to Moderate Symptoms and in Healthcare Workers With High Exposure Risk
Acronym: PREVENT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Concerned about the adverse effects of HCQ
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TCAI_PREVENT
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Symptomatic patients will be randomized to hydroxychloroquine (HCQ) vs no-HCQ group.
  Similarly, hospital staff with high risk of exposure will be randomized to HCQ vs no-HCQ group
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCQ arm (Active Comparator): COVID-19 positive cases will receive receive hydroxychloroquine sulfate 400 mg twice daily on the day of enrollment, then 200 mg twice daily for the next 4 days for a 5 day total course.
  Staff randomized to this group will receive HCQ sulfate 400 mg/week for 4 weeks
  Interventions: Drug: Hydroxychloroquine Sulfate
- No-HCQ arm (No Intervention): Will receive standard treatment as needed, but no HCQ

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — Patients will receive hydroxychloroquine sulfate 400 mg twice daily on the day of enrollment, then 200 mg twice daily for the next 4 days for a 5 day total course.
  Staff will receive HCQ sulfate 400mg/week for 4 weeks
  Arms: HCQ arm

SUMMARY:
Few studies have reported the efficacy of HCQ in reducing the viral load and improving the severity of symptoms in hospitalized COVID-19 cases with serious respiratory infection. However, the prophylactic benefits of HCQ has not been clearly defined yet.

DETAILED DESCRIPTION:
This study is designed to evaluate the prophylactic efficacy of HCQ in COVID-19 cases with mild to moderate symptoms and in the hospital staff engaged in attending infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age at the time of enrollment
* COVID-19 test positive patients with mild-moderate symptoms including fever >37.50 F
* Consecutive consenting staff at ICU, ER and COVID-19 unit that have never been diagnosed with COVID-19

Exclusion Criteria:

* Exclusion criteria:
* Hepatic cirrhosis or active hepatitis B or C
* Severe renal disease
* Hospitalized for severe symptoms of COVID-19 (ARDS), on mechanical ventilation or ECMO
* Contraindication to HCQ
* Using HCQ for some other condition (i.e. SLE, rheumatoid arthritis)
* Pregnant or breast feeding
* Known history of long QT syndrome (QTc >500 ms on electrocardiogram)
* Seizure disorder
* Body weight <50kg
* Psoriasis
* Unwilling to provide informed consent

Ages: 18 Months to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Time to reach normal body temperature | 1 month
  Time to reach normal body temperature (TNBT), ≤37.50 C
Development of COVID-19 symptoms during HCQ preventive therapy in staff | 1 month
  Development of fever and/or other symptoms of COVID-19 during the 1 month of the HCQ therapy

SECONDARY OUTCOMES:
COVID-19 test result at follow-up in patients | 6 days
  Viral RNA test results at day 6 will be compared between the HCQ vs no-HCQ group
Worsening of symptoms in COVID-19 patients | 1 month
  Worsening of symptoms in COVID-19 patients requiring artificial ventilation during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — St. David's Medical Center

IPD SHARING:
Plan to Share IPD: Undecided